CLINICAL TRIAL: NCT07234266
Title: Effect of Restorative Material Selection on Periodontal and Clinical Success in Teeth Restored With Indirect Restorations Fabricated by Additive Manufacturing After Deep Margin Elevation: A One-Year Clinical Follow-Up Study
Brief Title: The Effect of Material Choice on Clinical Outcomes in Deep Margin Elevation
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mersin University (Other)
Responsible Party: Principal Investigator, Esra Cengiz Yanardag, Professor, Mersin University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2025/909
Record Dates: First submitted 2025-11-14; First posted 2025-11-18 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Deep Marginal Elevation
Keywords: deep margin elevation; indirect restoration; additively manufactured; composite resin

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Saremco print resin- 3M Filtek One Bulk Fill Restorative (Active Comparator): The teeth is restored with Saremco print resin after deep margin elevation is performed with 3M Filtek One Bulk Fill Restorative.
  Interventions: Device: 3d printed resin restoration with deep margin elevation
- Saremco print resin- GC Gaeanial Universal Injectable (Active Comparator): The teeth is restored with Saremco print resin after deep margin elevation is performed with GC Gaeanial Universal Injectable
  Interventions: Device: 3d printed resin restoration with deep margin elevation
- Varseosmile TriniQ resin- 3M Filtek One Bulk Fill Restorative (Active Comparator): The teeth is restored with Varseosmile TriniQ resin after deep margin elevation is performed with 3M Filtek One Bulk Fill Restorative
  Interventions: Device: 3d printed resin restoration with deep margin elevation
- Varseosmile TriniQ resin- GC Gaeanial Universal Injectable (Active Comparator): The teeth is restored with Varseosmile TriniQ resin after deep margin elevation is performed with GC Gaeanial Universal Injectable
  Interventions: Device: 3d printed resin restoration with deep margin elevation

INTERVENTIONS:
Device: 3d printed resin restoration with deep margin elevation — The teeth are restored with 3D printed permanent resins after deep margin elevation

SUMMARY:
In dentistry, particularly in posterior teeth with extensive caries or old restorations, the extension of restoration margins below the gingival level presents a significant clinical challenge. In such cases, restorative procedures become more complicated, periodontal health may be adversely affected, and long-term tissue loss can occur. To overcome this problem, the "Deep Margin Elevation" technique has been developed. This approach aims to raise subgingival margins caused by caries or fractures above the gingival level, thereby providing a healthier and more favorable foundation for successful treatment.

In this study, two different materials will be used for deep margin elevation, followed by restoration of the teeth with indirect restorations fabricated using additive manufacturing technology, which has become increasingly popular in recent years. Two different additive manufacturing resins will also be applied in the restorative phase. The teeth treated with deep margin elevation and indirect restorations will be evaluated at baseline, 6 months, and 12 months according to the FDI criteria, as well as periodontal parameters due to the involvement of the gingival region.

This study aims to highlight the importance of material selection in restorative treatment planning and to scientifically demonstrate the impact of the applied technique on surrounding tissues. Furthermore, it will provide an evidence-based perspective on how adopting a tissue-friendly approach during restorative procedures may contribute to favorable long-term outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Patients who apply to Mersin University Faculty of Dentistry between 01.12.2025 and 01.03.2026 for restorative treatment of their teeth
* Patients aged between 18 and 84 years
* Patients without parafunctional habits (such as bruxism, clenching, or foreign object chewing)
* Vital or non-vital molar and premolar teeth with a clinical indication for inlay/onlay restoration
* Teeth with deep cavities and margins located at or slightly below the gingival level
* Defects limited to the occlusal surface and one proximal surface
* Occlusal defects extending beyond one-third of the distance between fissure and cusp tip, including at least one cusp
* Posterior teeth with an indication for deep margin elevation without violation of the biologic width
* Teeth with opposing natural teeth or fixed prosthetic restorations
* Teeth with the presence of adjacent proximal contacts

Exclusion Criteria:

* Teeth with fractures or cracks
* Patients with temporomandibular joint disorders
* Patients with malocclusion, bruxism, or parafunctional habits
* Posterior teeth without opposing natural teeth or fixed prosthetic restorations
* Posterior teeth without adjacent proximal contacts
* Patients with a history of allergy to the components of the restorative materials used
* Patients with severe gingival enlargement, gingival recession, or active periodontal disease
* Teeth requiring deep margin elevation that present with non-physiological mobility, fistula, or periapical lesions

Ages: 18 Years to 84 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2026-06 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Clinical performance and periodontal paremetres | Baseline, 6 months, 12 months
  The clinical evaluation of restorations bonded to teeth will be performed using World Dental Federation (FDI) criteria in addition to periodontal parameters. Regarding FDI criteria, each property is typically scored on a 1 to 5 scale: 1- Clinically excellent, 2- Clinically good, 3- Clinically sufficient, 4- Clinically insufficient, 5- Clinically poor Regarding gingival index, 0-1: Clinically acceptable, 1-2: Clinically unacceptable Regarding plaque index, 0-1 clinically acceptable, 2 borderline, 3 clinically unacceptable In terms of probing pocket depth, ≤3 mm clinically acceptable, 4-5 mm borderline ≥6 mm s clinically unacceptable

CONTACTS AND LOCATIONS:
Locations (1):
- Mersin University, Faculty of Dentistry, Mersin, Mersin, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided